CLINICAL TRIAL: NCT00206947
Title: PHARMACOLOGICAL TREATMENT OF COGNITIVE DEFICITS IN SCHIZOPHRENIC PATIENTS: The Effects of Central Cholinergic Augmentation on Cognitive Deficits and Psychopathology
Brief Title: The CAMPUS Project: Cholinergic Augmentation of Cognitive Deficits in Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No more funding
Sponsor: Birte Glenthoj (Other)
Collaborators: Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Birte Glenthoj, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 363051; KF 02-033/02; DMA 2612-2013
Record Dates: First submitted 2005-09-11; First posted 2005-09-21 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
Keywords: Cognitive deficits; Cholinergic Augmentation; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Donepezil; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: donepezil (5-10 mg/day)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil (5-10 mg/day) — Donepezil will be administered in a dose optimized for treatment, to patients who are stabilized on a ziprasidone treatment
  Other Names: Aricept, Zeldox
  Arms: 1
Drug: Placebo — Placebo will be added to the medication of schizophrenia patients who are first stabilized on a ziprasidone treatment
  Other Names: Zeldox
  Arms: 2

SUMMARY:
The present study will specify and delineate the separate components of cognitive deficits and examine the effects of adjunctive cholinergic augmentation on these cognitive deficits as well as psychopathology in schizophrenic patients treated with an antipsychotic compound with no aberrant binding affinity for the cholinergic receptor system. The hypothesis is that cholinergic augmentation using donepezil will improve cognitive deficits, sensory gating deficits, and psychopathology in schizophrenic patients treated with an atypical antipsychotic (ziprasidone).

DETAILED DESCRIPTION:
The purpose of the study was to examine the effects of cholinergic augmentation of atypical antipsychotic medication on:

* Cognitive deficits
* Sensorimotor gating
* Psychopathology

The primary objective was to examine:

• The effects of donepezil, compared to the effects of placebo, on cognitive function, sensorimotor gating and psychopathology in patients treated with an atypical antipsychotic (ziprasidone).

Secondary objectives are to examine:

* The effect of donepezil, compared to the effects of placebo, on cognitive function, sensorimotor gating and psychopathology in patients treated with ziprasidone.
* Which specific areas of cognitive deficits benefit from cholinergic augmentation of atypical antipsychotic treatment.
* The interactions between cognitive deficits and psychopathology: To what extent the effects of cholinergic augmentation on psychopathology, sensorimotor gating, and cognition are independent or correlated.
* Which specific brain areas are activated during cholinergic augmentation of treatment with an atypical antipsychotic drug (ziprasidone).

Participants: Schizophrenic men and women between the ages 18 to 55 who meet the ICD-10 criteria for schizophrenia living in the catchment area of the psychiatric departments of Bispebjerg University Hospital,Rigshospitalet, or Psychiatric Center, Glostrup. Patients can be either unmedicated, or need to be switched from other antipsychotic medications due to side-effects, or lack of effect on negative symptoms, positive symptoms, or cognitive function. Patients can be enrolled in the study as inpatients or outpatients, and changes in hospitalization status during the trial are allowed. Patients were stabilized on antipsychotic medication (ziprasidone) before they were randomized to treatment with either donepezil or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Men and women between the ages 18 to 55 who meet the ICD-10 criteria for schizophrenia living in the catchment area of the psychiatric departments of Bispebjerg University Hospital, Psychiatric Center, Glostrup and Rigshospitalet. Patients can be either unmedicated, or need to be switched from other antipsychotic medications due to side-effects, or lack of effect on negative symptoms, positive symptoms, or cognitive function.
* Controls: Healthy men and women matched according to gender, age, and socio-economic status (determined by the level of education and income of parents).

Exclusion Criteria:

* Patients: Patients hospitalized against their will. Patients with a serious medical illness or with laboratory abnormalities, where pharmacotherapy poses a substantial clinical risk; pregnant or lactating patients; patients with organic psychosis, a history of severe head trauma or convulsive disorders, or patients with mental retardation. Patients with significant alcohol- or drug dependence are excluded.
* Controls: Pregnant or lactating women; a history of severe head trauma; mental retardation; learning difficulties; a history of psychiatric illness or a familial predisposition to psychiatric illness (in first-degree relatives); significant alcohol- or drug dependence; episodic incidents of excessive alcohol consumption or drug abuse are not reasons for exclusion. Abuse is monitored by interviewing patients and by measuring the urine content for amphetamine, cannabinoles, opiates, and benzodiazepines. Concomitant use of benzodiazepines for agitation or insomnia (oxazepam up to 45 mg daily) is allowed when needed and when used conservatively during the trial. Use of anticholinergic compounds is not allowed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2002-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
PANSS (Positive and Negative Symptom Scale) | baseline and after treatment
the CGI (Clinical Global Impression scale) | baseline and after treatment
the ESRS (Extrapyramidal Symptom Rating Scale) | baseline and after treatment
Cognitive functions: A comprehensive test battery focuses on central cognitive deficits in schizophrenia: i.e. memory functions, attention, executive functions, reaction time, as well as pre-morbid and current intelligence. | baseline and after treatment

SECONDARY OUTCOMES:
MRI | baseline and after treatment
fMRI | baseline and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Birte Glenthoj, MD, DMSc., Study Director — Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Psychaitric Center Glostrup, Ndr. Ringvej, DK-2600 Glostrup, Denmark
Locations (4):
- Denmark (4):
  - Dept. of Psychiatry O, Rigshospitalet, Blegdamsvej 9, Copenhagen
  - Center for Neuropsychiatric Schizophrenia Research, University of Copenhagen, Dept. F, Bispebjerg Hospital, Copenhagen NV
  - Psychiatric Center, Glostrup, Glostrup Municipality
  - Danish Research Center for Magnetic Resonance Imaging, Hvidovre Hospital, Hvidovre

REFERENCES:
- See also: Center for Neuropsychiatric Schizophrenia Research (CNSR) — http://www.cnsr.dk